CLINICAL TRIAL: NCT03137004
Title: A Single-arm Phase II Trial of Biweekly Docetaxel and S-1 Combination Therapy as Second-line Treatment for Advanced Gastric Cancer
Brief Title: Docetaxel and S-1 Combination Therapy as Second-line Treatment for Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FNF-005
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Advanced Gastric Cancer
MeSH Terms: interventions — Docetaxel; S 1 (combination); titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- biweekly DS (Experimental): The biweekly DS regimen consisted of Docetaxel (50mg/m2) and S-1 (40mg/m2)
  Interventions: Drug: Docetaxel; Drug: S-1

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 50mg/m2 in 60 min on day 1 and repeated every 14 days.
  Other Names: Taxotere
Drug: S-1 — S-1 was administered orally at 40 mg/m2 twice daily on days 1-7 of each cycle. Patients with a body surface area of less than 1.25 m2 received 80 mg S-1 daily, those with a body surface area of 1.25 m2 or more but less than 1.5 m2 received 100 mg S-1 daily, and those with a body surface area of 1.5 m2 or more received 120 mg S-1 daily.
  Other Names: TS-1

SUMMARY:
A single-arm phase II study to evaluate the efficacy and safety of docetaxel plus S-1 (DS) as second-line treatment in patients with AGC.

DETAILED DESCRIPTION:
For patients with advanced gastric cancer, combination chemotherapy has been shown to improve the quality of life and overall survival (OS) compared with best supportive care alone. Docetaxel is an active agent for treating patients with gastric cancer. S-1, an oral 5-FU prodrug, is active against AGC as a single agent or in combination with cisplatin in phase III trials. Therefore, a single-arm phase II study was conducted to investigate the efficacy and safety of biweekly docetaxel and S-1 (DS) combination therapy as second-line treatment in patients with previously treated advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old;
2. Histologically or cytologically confirmed unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma;
3. The patient has experienced disease progression during treatment or within 4 months after the last dose of first-line therapy without taxanes for metastatic disease.
4. Relapse within 6 months after adjuvant chemotherapy;
5. ECOG (Eastern Cooperative Oncology Group)performance status 0-2;
6. At least 1 measurable lesion should be present（RECIST1.1）
7. Available Organ function: Neutrophils>2g/L, Hemoglobin>9g/L, Blood platelet >100g/L; Alanine aminotransferase(ALT） and Aspartate aminotransferase(AST)<1.5 ULN(upper limit of normal); Total bilirubin(TBIL)<1.0 ULN; Cr <1.0ULN
8. Signed informed consent.
9. Life expectancy ≥3 months;

Exclusion Criteria:

1. Previous treatment with taxanes (not including intraperitoneal use of taxanes);
2. Known history of hypersensitivity to study drugs;
3. Active CNS metastases not controllable with radiotherapy or corticosteroids;
4. Pregnant or breast feeding women;
5. Severe co-morbid illness and/or active infections;
6. Active and uncontrollable bleeding from gastrointestinal tract
7. Patients receiving a concomitant treatment with drugs interacting with S-1 such as flucytosine, phenytoin, or allopurinol;
8. Other co-existing malignancies or malignancies diagnosed within the last 5 years(except cured cutaneum carcinoma or carcinoma in situs of cervix);
9. Known HIV infecton.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2018-04-10 (Estimated); Study Completion 2018-10-10 (Estimated)

PRIMARY OUTCOMES:
six-month overall survival | 6 months

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 6 months
Overall Survival (OS) | 12 months
Progression-Free Survival (PFS) | 12 months
Adverse Event（AE） | NCI CTC 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Rongbo Lin, MD, Study Chair — Fujian Cancer Hospital
Locations (1):
- Rongbo Lin, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No